CLINICAL TRIAL: NCT03195166
Title: Hemodynamic Effects of Continuous Spinal Anesthesia in Patient Aged Over 65 Years Undergoing Total Knee Arthroplasty
Brief Title: Hemodynamic Effects of Continuous Spinal Anesthesia in Patient Aged Over 65 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, professor, University Tunis El Manar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101/2017
Record Dates: First submitted 2017-06-04; First posted 2017-06-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hemodynamic Instability
Keywords: elderly spinal anesthesia

STUDY DESIGN:
Intervention Model Description: The aim of this study was to investigate the hemodynamic effects of continuous spinal anesthesia in elderly patients. An oral intake of 250 ml of water was taken 2 hours before surgery.
  Radial arterial catheter was putted under local anesthesia and connected to the FloTrac sensor/Vigileo haemodynamic monitoring system.
  Fluid therapy was limited to 4 ml/kg/h until tourniquet release.
  Subarachnoid puncture was performed at the L3-S1 interspace. An initial dose of 2,5 mg isobaric 0,5% bupivacaine was injected. Additional 2,5 mg isobaric 0,5% bupivacaine doses were injected every 10 minutes until sensory blockade reached T10.
  Ephedrine 6 to 9 mg was given if systolic arterial pressure < 90 mmHg. Investigators measured blood pressure (systolic, diastolic and mean), stroke volume and cardiac output every 5 minutes from beginning of the operation and until 2 hours after the end.
  Number of hypotension episodes and ephedrine consumption were noted.
Masking Description: consecutive patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hemodynamic profile (Experimental): FloTrac sensor/Vigileo
  Interventions: Diagnostic Test: FloTrac sensor/Vigileo

INTERVENTIONS:
Diagnostic Test: FloTrac sensor/Vigileo — blood pressure (systolic, diastolic and mean), stroke volume cardiac output ephedrine consumption after bupivacaine continuous spinal anesthesia

SUMMARY:
Compared to single-dose spinal anesthesia, continuous spinal anesthesia using small titrated doses of local anesthetic, was safe, efficient and provided better hemodynamic profile in elderly patients.

The aim of this study was to investigate the hemodynamic effects of continuous spinal anesthesia in elderly patients undergoing knee arthroplasty.

Investigators use the FloTrac sensor/Vigileo haemodynamic monitoring system to assess modification blood pressure, stroke volume and cardiac output during anesthesia and specialy after every bolus of spinal anesthesia, after inflating the tourniquet and after putting it off.

they recorded number of hypotension episodes, ephedrine bolus and consumption until 2 hours after the end of surgery.

DETAILED DESCRIPTION:
The aim of this study was to investigate the hemodynamic effects of continuous spinal anesthesia (CSA) in elderly patients undergoing knee arthroplasty.

Inclusion criteria:

Adult patients, aged more than 65 years scheduled for elective total knee arthroplasty under regional anesthesia.

Study Design :

Patients had a transthoracic echocardiography one to three months before the surgical procedure, performed by a cardiologist.

An oral intake of 250 ml of water was taken 2 hours before surgery. In the operating room, patients received monitoring with electrocardiogram, pulse oximetry and had their blood pressure measured and recorded via an indwelling radial arterial catheter putting under local anesthesia.

This catheter was connected to the FloTrac sensor/Vigileo haemodynamic monitoring systeme to track continuously stroke volume and cardiac output.

All patients were given nasal oxygen during all the procedure to keep oxygen saturation > 95 %. Fluid therapy was limited to 4 ml/kg/h until tourniquet release.

Subarachnoid puncture was performed with a 19-Gauge Tuohy needle at the L3-S1 interspace using a midline approach. Three cm of a 22-Gauge catheter was introduced through the needle. An initial dose of 2,5 mg isobaric 0,5% bupivacaine was injected through the catheter. Additional 2,5 mg isobaric 0,5% bupivacaine doses were injected every 10 minutes until sensory blockade reached T10.

Ephedrine 6 to 9 mg was given if systolic arterial pressure < 90 mmHg or < 100 mmHg with clinical signs of poor tolerance (dizziness, anxiety, dyspnea, vomiting).

Sample size We included 20 patients in this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged more than 65 years
* scheduled for elective total knee arthroplasty
* under regional anesthesia

Exclusion Criteria:

* contraindication to regional anesthesia
* or the patients who refused to give consent,
* patients with anemia (hemoglobin < 13 g/dl for male and hemoglobin < 12 g/dl for female),
* cardiac arrhythmias,
* NYHA score > 2,
* ASA > 2
* Cardiac ejection fraction < 50 %,
* valvulopathy,
* pulmonary artery hypertension
* and relaxation abnormality

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
hemodynamic profile during continuous spinal anesthesia in elderly | Day 0
  cardiac output , L/min

SECONDARY OUTCOMES:
blood pressure variation | Day 0
  systolic blood pressure, diastolic blood pressure, mean blood pressure, mmHg
ephedrine use | Day 0
  ephedrine consumption , mg
stoke volume modification | Day 0
  stroke volume, L

CONTACTS AND LOCATIONS:
Overall Officials: KAABACHI OLFA, PROF, Study Chair — KASSAB ORTHOPEDIC INSTITUTE
Locations (1):
- Kassab orthopedic Institute, Tunis, La Manouba, Tunisia

IPD SHARING:
Plan to Share IPD: No